CLINICAL TRIAL: NCT00525239
Title: HIV Antiretroviral Drugs and Metabolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Carl Grunfeld, M.D., Ph.D., Principal Investigator, Northern California Institute for Rerseach and Education
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: DK66999
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: HIV Infections
Keywords: Lipids; lipoproteins; VLDL; triglycerides; apo B100; HDL; apo A1; endothelial dysfunction; insulin secretion; hyperglycemic clamp; HIV-seronegative Volunteers; HIV-infected subjects starting an efavirenz-based regimen; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; Lopinavir; atazanavir, ritonavir drug combination; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1: Ritonaivr (Experimental): Pre and post ritonavir, lopinavir/ritonavir or atazanavir/ritonavir
  Interventions: Drug: ritonavir, lopinavir/ritonavir, atazanavir/ritonavir, efavirenz

INTERVENTIONS:
Drug: ritonavir, lopinavir/ritonavir, atazanavir/ritonavir, efavirenz — 100 mg, twice daily, for four weeks

SUMMARY:
Hypothesis 1: Ritonavir-based regimens increase triglycerides and VLDL by both increasing VLDL production and decreasing VLDL clearance.

Specific Aim 1A: To quantify the effect of ritonavir on VLDL production and clearance using stable isotope turnover and other clearance methods.

Specific Aim 1B: To determine the composition of the triglyceride rich particles.

Protocol 1: The effects of ritonavir-based regimens on VLDL production, VLDL clearance and triglyceride-rich lipoprotein composition in healthy normal volunteers. HIV-seronegative volunteers will be studied before and at the end of four weeks of taking ritonavir, lopinavir/ritonavir or atazanavir/ritonavir.

Hypothesis 2: NNRTI drugs do not increase HDL by increasing apo AI production, but rather by decreasing apo AI clearance, prolonging time in circulation.

Specific Aim 2A: To determine the composition of HDL before and after NNRTI and assess its function.

Specific Aim 2B: To quantify the effect of NNRTI on apo AI production and clearance using stable isotopes.

Specific Aim 2C: To determine if the NNRTI induced increase in HDL is accompanied by improvement in flow mediated vasodilation and circulating markers of endothelial function Protocol 2A: The effects of efavirenz on HDL composition, HDL function, apo AI production, apo AI clearance, flow mediated vasodilation and circulating markers of endothelial dysfunction in healthy normal volunteers. HIV-seronegative volunteers will be studied before and at the end of six weeks of taking efavirenz.

Protocol 2B: The effects of starting an efavirenz-based regimen on HDL composition, HDL function, apo AI production, apo AI clearance, flow mediated vasodilation and circulating markers of endothelial dysfunction in patients with HIV infection. HIV-infected patients whose care providers have prescribed an efavirenz-based regimen will be studied before and after six weeks of starting efavirenz.

Hypothesis 3: Ritonavir-based PI regimens impair insulin secretion. Specific Aim 3: To determine which ritonavir-based PI regimens alter insulin secretion.

Protocol 3: The effects of ritonavir-based regimens on insulin secretion in healthy normal volunteers. HIV-seronegative volunteers will be studied before and at the end of four weeks of taking ritonavir, lopinavir/ritonavir or atazanavir/ritonavir.

ELIGIBILITY:
Inclusion Criteria:

Protocols 1, 2A and 3 HIV negative, healthy normal volunteers, age > 18 years old.

Protocol 2B HIV-infected subjects, age > 18 years old and documented to have HIV-1 infection for ≥ 6 months, being started on efavirenz by their health care provider.

Exclusion Criteria:

Protocols 1, 2A and 3 Coronary artery disease, peripheral vascular disease, impaired fasting glucose (glucose > 100 mg/dl), obese (BMI > 30), dyslipidemia (triglycerides > 190 mg/dl, LDL-C > 190), anemia (Hct < 39), hypertension (BP> 140/90 mmHg or on medication), blood pressure <100 mmHg, renal disease (creatinine > 1.6), LFT > ULN, or use within 30 days of systemic glucocorticoids, anabolic steroids, growth hormone, niacin, antipsychotics, or lipid lowering medications. Women will be tested for pregnancy immediately prior to each inpatient study and excluded if pregnant. For Specific Aim 2, additional exclusion criteria include history of depression requiring treatment, psychosis, hallucinations or delusions; use of cGMP specific phosphodiesterase 5 inhibitors (e.g., sildenafil) within 7 days of study; or history of adverse reaction to nitrates.

Protocols 1, 2A and 3 Currently on an NNRTI, coronary artery disease, peripheral vascular disease, recent opportunistic infection (within two months), impaired fasting glucose (glucose > 100 mg/dl) or diabetes, anemia (Hct < 39), hypertension (BP > 140/90 mmHg or on medication), blood pressure <100 mmHg, renal disease (Creatinine > 1.6), LFT > 2x ULN, use of cGMP specific phosphodiesterase 5 inhibitors (e.g., sildenafil) within 7 days of study, history of adverse reaction to nitrates, use within 30 days of anabolic steroids, systemic glucocorticoids, growth hormone, niacin, antipsychotics, or lipid lowering medications. Women will be tested for pregnancy immediately prior to each inpatient study and excluded if pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-03; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Effect of HIV Protease Inhibitors on Glucose Metabolism by Hyperglycemic Clamp | 4 weeks

SECONDARY OUTCOMES:
Effect of HIV Protease Inhibitors on Oral Glucose Tolerance Test | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carl Grunfeld, M.D., Ph.D., Principal Investigator — Northern California Institute for Research and Education
Locations (1):
- Department of Veterans Affairs Medical Center, San Francisco, California, United States

REFERENCES:
- [Result] Noor MA, Lo JC, Mulligan K, Schwarz JM, Halvorsen RA, Schambelan M, Grunfeld C. Metabolic effects of indinavir in healthy HIV-seronegative men. AIDS. 2001 May 4;15(7):F11-8. doi: 10.1097/00002030-200105040-00001. PMID 11399973
- [Result] Noor MA, Seneviratne T, Aweeka FT, Lo JC, Schwarz JM, Mulligan K, Schambelan M, Grunfeld C. Indinavir acutely inhibits insulin-stimulated glucose disposal in humans: a randomized, placebo-controlled study. AIDS. 2002 Mar 29;16(5):F1-8. doi: 10.1097/00002030-200203290-00002. PMID 11964551
- [Result] Lee GA, Seneviratne T, Noor MA, Lo JC, Schwarz JM, Aweeka FT, Mulligan K, Schambelan M, Grunfeld C. The metabolic effects of lopinavir/ritonavir in HIV-negative men. AIDS. 2004 Mar 5;18(4):641-9. doi: 10.1097/00002030-200403050-00008. PMID 15090769
- [Result] Lee GA, Mafong DD, Noor MA, Lo JC, Mulligan K, Schwarz JM, Schambelan M, Grunfeld C. HIV protease inhibitors increase adiponectin levels in HIV-negative men. J Acquir Immune Defic Syndr. 2004 May 1;36(1):645-7. doi: 10.1097/00126334-200405010-00017. No abstract available. PMID 15097312
- [Result] Schwarz JM, Lee GA, Park S, Noor MA, Lee J, Wen M, Lo JC, Mulligan K, Schambelan M, Grunfeld C. Indinavir increases glucose production in healthy HIV-negative men. AIDS. 2004 Sep 3;18(13):1852-4. doi: 10.1097/00002030-200409030-00017. PMID 15316349
- [Result] Lee GA, Rao MN, Grunfeld C. The effects of HIV protease inhibitors on carbohydrate and lipid metabolism. Curr HIV/AIDS Rep. 2005 Feb;2(1):39-50. doi: 10.1007/s11904-996-0008-z. PMID 16091248
- [Result] Lee GA, Lo JC, Aweeka F, Schwarz JM, Mulligan K, Schambelan M, Grunfeld C. Single-dose lopinavir-ritonavir acutely inhibits insulin-mediated glucose disposal in healthy volunteers. Clin Infect Dis. 2006 Sep 1;43(5):658-60. doi: 10.1086/505974. Epub 2006 Jul 26. PMID 16886163
- [Result] Lee GA, Rao M, Mulligan K, Lo JC, Aweeka F, Schwarz JM, Schambelan M, Grunfeld C. Effects of ritonavir and amprenavir on insulin sensitivity in healthy volunteers. AIDS. 2007 Oct 18;21(16):2183-90. doi: 10.1097/QAD.0b013e32826fbc54. PMID 18090045
- [Derived] Taylor SA, Lee GA, Pao VY, Anthonypillai J, Aweeka FT, Schwarz JM, Mulligan K, Schambelan M, Grunfeld C. Boosting dose ritonavir does not alter peripheral insulin sensitivity in healthy HIV-seronegative volunteers. J Acquir Immune Defic Syndr. 2010 Nov;55(3):361-4. doi: 10.1097/QAI.0b013e3181e6a7d9. PMID 20595906
- [Derived] Pao VY, Lee GA, Taylor S, Aweeka FT, Schwarz JM, Mulligan K, Schambelan M, Grunfeld C. The protease inhibitor combination lopinavir/ritonavir does not decrease insulin secretion in healthy, HIV-seronegative volunteers. AIDS. 2010 Jan 16;24(2):265-70. doi: 10.1097/QAD.0b013e328333af1c. PMID 19890203